CLINICAL TRIAL: NCT05438407
Title: An Open-label, Single Arm Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of Leniolisib in Pediatric Patients Aged 4 to 11 Years With Activated Phosphoinositide 3-Kinase Delta Syndrome Followed by an Open-label Long-term Extension
Brief Title: Pediatric Patients Aged 4 to 11 Years With APDS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pharming Technologies B.V. (Industry)
Collaborators: CMIC Co, Ltd. Japan (Industry); Labcorp Central Laboratory (Unknown); Fortrea (Industry); Aixial Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LE 3301
Record Dates: First submitted 2022-05-20; First posted 2022-06-30 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: APDS
MeSH Terms: interventions — leniolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Leniolisib (Experimental): Leniolisib - Film Coated Tablets Leniolisib tablets in 10 and 30 mg strengths administered orally BID by body weight for 12 weeks for Part I and for 1 year for Part II.
  Interventions: Drug: Leniolisib

INTERVENTIONS:
Drug: Leniolisib — The doses selected range from 20 to 70 mg BID (resulting in total daily doses ranging from 40 to 140 mg per day) based on weight. The doses will be administered as (a combination of) 10 mg and 30 mg tablets

SUMMARY:
This is a 2-part, prospective, open-label, single arm, multicenter study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PDx), and efficacy of leniolisib in at least 15 pediatric patients (aged 4 to 11 years) with activated phosphoinositide 3-kinase delta (PI3Kδ) syndrome (APDS).

DETAILED DESCRIPTION:
Part I will consist of a 12-week period to assess the safety and efficacy of treatment with leniolisib. Part II will consist of a 1-year, long-term, safety follow-up extension with a possible interim analysis.

The leniolisib doses to be used in study were selected based on safety, tolerability, PK, and PDx data from the adult Phase 2/3 study, as well as PK modeling data. In both parts of the study, leniolisib will be administered orally based on weight.

ELIGIBILITY:
Diagnosis and main criteria for inclusion and exclusion:

Patients must satisfy all of the following criteria at the screening visit unless otherwise stated:

1. Patient is male or female and between the age of 4 to 11 years old at the time of the first study procedure.
2. Patient weighs ≥13 kg and <45 kg at baseline.
3. Patient has a confirmed PI3Kδ genetic mutation of either the PIK3CD (APDS1) or PIK3R1 (APDS2) gene.
4. Patient has at least 1 measurable nodal lesion on magnetic resonance imaging/low-dose computed tomography within 6 months of screening.
5. Patient has nodal or extranodal lymphoproliferation and clinical findings consistent with APDS (eg, a history of repeated oto-sino-pulmonary infections and/or organ dysfunction consistent with APDS).
6. Patient has the ability to ingest unaltered study-related medications without difficulty in the investigator's opinion.
7. At screening, vital signs (systolic blood pressure [BP], diastolic BP, and pulse rate) will be assessed in the sitting position after the patient has been at rest for at least 3 minutes. Patient's sitting vital signs should be within the following ranges:

   * Systolic BP: Less than the 95th percentile adjusted for sex, age, and height percentile.
   * Diastolic BP: Less than the 95th percentile adjusted for sex, age, and height percentile.
   * Heart rate (HR):

     i) Age 4 to <10 years: 60 to 140 bpm ii) Age ≥10 years: 50 to 100 bpm
8. Institutional review board-/independent ethics committee-approved written informed consent/assent and privacy language as per national and local regulations must be obtained from the patient and parent/legal guardian prior to any study-related procedures.
9. Patient parent/legal guardian is willing and able to complete the informed consent/assent process and comply with study procedures and visit schedule.
10. Patient parent/legal guardian agrees patient will not participate in any other interventional study while enrolled in this study.
11. Female patients should be of non-childbearing potential at screening (should not have reached menarche). Male patients with partners of childbearing potential should be willing to use a highly effective method of contraception for at least 30 days after the last study procedure if at risk of pregnancy.
12. Female patient and parent/legal guardian must agree to the following if menses develops after screening, up to 30 days after the last study procedure:

    * True sexual abstinence defined as refraining from heterosexual activity during the entire period of the study through 6 months post-study or
    * Using a highly effective method of contraception for at least 30 days after the last study procedure if at risk of pregnancy.

Patients will be excluded from the study if they satisfy any of the following criteria at the screening visit unless otherwise stated:

1. Patient has previous or concurrent use of immunosuppressive medication such as:

   a. An mTOR inhibitor (eg, sirolimus, rapamycin, everolimus) or a PI3Kδ inhibitor (selective or non-selective PI3K inhibitors) within 6 weeks prior to first dose.

   i. Short-term use for up to a total of 5 days is allowed but only up to 1 month prior to enrollment in the study.

   b. B cell depleters (eg, rituximab) within 6 months prior to first dose of study medication.

   i. If patient has received prior treatment with a B cell depleter, absolute B lymphocyte counts in the blood must have regained normal values.

   c. Belimumab or cyclophosphamide within 6 months prior to first dose of study medication.

   d. Cyclosporine A, mycophenolate, 6-mercaptopurine, azathioprine, or methotrexate within 3 months prior to first dose of study medication.

   e. Systemic glucocorticoids above a dose equivalent to either ≥2 mg/kg of body weight or ≥20 mg/day of prednisone/prednisolone or equivalent.

   f. Other immunosuppressive medication where effects are expected to persist at start of dosing of study medication.
2. Patient has a history or current diagnosis of electrocardiogram (ECG) abnormalities indicating significant risk of safety for patients participating in the study such as:

   1. History of familial long QT syndrome or known family history of Torsades de Pointes.
   2. Concomitant clinically significant cardiac arrhythmias (eg, sustained ventricular tachycardia, and clinically significant second or third degree atrioventricular block without a pacemaker).
   3. Resting QTc (Fridericia preferred, but Bazett acceptable) >460 msec if the measurement is confirmed with an additional ECG repeated as soon as possible.
   4. Concomitant use of agents known to prolong the QT interval unless it can be permanently discontinued for the duration of the study.
3. Patient is currently using a medication known to be a strong inhibitor or moderate or strong inducer of isoenzyme cytochrome P450 (CYP)3A, if treatment cannot be discontinued or switched to a different medication prior to starting study treatment.
4. Patient is currently using medications that are metabolized by isoenzyme CYP1A2 and have a narrow therapeutic index (drugs whose exposure-response indicates that increases in their exposure levels by the concomitant use of potent inhibitors may lead to serious safety concerns [eg, Torsades de Pointes]).
5. Patient had been administered live vaccines (this includes any attenuated live vaccines) starting from 6 weeks before the anticipated first study drug administration, during the study, and up to 7 days after the last dose of leniolisib.
6. Patient has clinically significant abnormalities in hematology or clinical chemistry (blood chemistry or urinalysis) parameters as determined by the investigator or medical monitor.
7. Patient has liver disease or liver injury as indicated by clinically significant abnormal liver function tests (alanine aminotransferase and aspartate aminotransferase >2.5 times upper limit of normal), history of renal injury/renal disease (eg, renal trauma, glomerulonephritis, or one kidney only), or presence of impaired renal function as indicated by a serum creatinine level >1.5 mg/dL (133 μmol/L).
8. Patient has moderate or severe hepatic impairment (Child-Pugh Class B or C).
9. Patient is receiving concurrent treatment with another investigational therapy or use of another investigational therapy less than 4 weeks from the first study procedure.
10. Patient has active hepatitis B (eg, hepatitis B surface antigen reactive) or active hepatitis C (eg, hepatitis C virus RNA [qualitative] is detected) at screening.
11. Patient has human immunodeficiency virus (HIV) infection (HIV 1 or 2) at screening.
12. Patient has a positive coronavirus disease 19 result (polymerase chain reaction or antigen) within 1 week prior to first dose. The patient can be rescreened after a subsequent negative result.
13. Patient has a history of malignancy (except lymphoma) within 3 years before the first study procedure or has evidence of residual disease from a previously diagnosed malignancy.
14. Patient has a previous diagnosis of lymphoma that has been treated with chemotherapy, radiotherapy, or transplant within 1 year of the first study procedure or is anticipated to require lymphoma treatment within 6 months of the first study procedure.
15. Patient has a history of uncontrolled diabetes mellitus within 3 months of the first study procedure.
16. Patient has had major surgery requiring hospitalization or radiotherapy within 4 weeks prior to the first study procedure.
17. Patient has uncontrolled chronic or recurrent infectious disease (with the exception of those that are considered to be characteristic of APDS) or evidence of tuberculosis infection as defined by a positive Mantoux tuberculin skin test at screening. If presence of latent tuberculosis is established, then treatment according to local country guidelines must have been completed before patients can be considered for enrollment.
18. Patient has a known allergy or history of hypersensitivity to study defined medications or any ingredients of the medications, including the following common excipients:

    * Lactose monohydrate
    * Microcrystalline cellulose
    * Sodium starch glycolate (Type A)
    * Hypromellose
    * Magnesium stearate
    * Colloidal silicon dioxide
    * Opadry yellow
19. Patient has a planned or expected major surgical procedure.
20. Patient or parent/legal guardian is unable or unwilling to comply with study procedures or is unable to travel for repeat visits.
21. Patient or parent/legal guardian is unwilling to keep study results/observations confidential or to refrain from posting confidential study results/observations on social media sites.
22. Patient or parent/legal guardian refuses to sign consent/assent form.
23. Patient has other underlying medical condition that, in the opinion of the investigator, would impair the ability of the patient to receive or tolerate the planned procedures or follow-up.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Part I & II: Number of Participants with Treatment-emergent adverse events (TEAEs), Serious Adverse Events (SAEs) , and Adverse Events (AEs) | From baseline to end of 12 weeks, & From baseline to through study completion, an average of 1 year, plus 30 days
  Number of Participants with TEAEs, SAEs, and AEs leading to discontinuation of study drug
Part I & II: Change from baseline in clinical laboratory test results | From baseline to end of 12 weeks, & From baseline to through study completion, an average of 1 year
  Number of Participants with change in clinical laboratory test results (hematology, blood chemistry, urinalysis)
Part I & II: Change from baseline in vital signs | From baseline to end of 12 weeks, & From baseline to through study completion, an average of 1 year
  Number of Participants with change in vital signs
Part I & II: Change from baseline in physical examination findings | From baseline to end of 12 weeks, & From baseline to through study completion, an average of 1 year
  Number of Participants with change in physical examination findings
Part I & II: Change from baseline in electrocardiograms (ECGs) | From baseline to end of 12 weeks, & From baseline to through study completion, an average of 1 year, plus 30 Days
  Number of Participants with change in electrocardiograms (ECGs)
Part I & II: Change from baseline in growth and physical development | From baseline to end of 12 weeks, & From baseline to through study completion, an average of 1 year
  Number of Participants with change in growth and physical development
Part I & II: Reduction in lymphoproliferation as measured by MRI or low-dose CT | Part I: Baseline and Day 85 Part II: at Day 252, through study completion, an average of 1 year
  For the assessment of the impact of leniolisib on lymphoproliferation, patients will be scanned in an MRI or a CT scanner as based on clinical practice and local regulation. Index lesions will be selected from measurable nodal and extra nodal lesions as per the Cheson methodology. The same imaging modality will be used throughout the study for the same patient. Patients will be assessed by MRI, or in sites where local practice and local authorities/IECs/IRBs approve CT scans for research purposes using a low-dose CT scan.
Part I: A Percentage of Inhibition of Unstimulated and Stimulated pAkt Levels in B Cells | Part I: Baseline, Days 29, 57 and 85
  The PDx effect of leniolisib will be assessed using ex vivo stimulated and unstimulated phosphorylation of Akt in B cells. Akt is a direct downstream target of activated PI3Kδ. Determination of the percentage (%) of CD20+ pAkt positive cells after ex vivo stimulation of whole blood is performed by flow cytometry analysis. Unstimulated cells will serve as controls.

SECONDARY OUTCOMES:
Part I: To evaluate changes in Pharmacokinetic (PK) profile/parameters | From baseline to end of 12 weeks of treatment]
  To evaluate changes in Cmax, Tmax AUC, T1/2
Part I: To evaluate changes in Pharmacodynamic (PD) profile/parameters | From baseline to end of 12 weeks of treatment]
  To evaluate changes in pAkt and Serum Immunoglobulin Profile
Part I: To assess the total drug exposure (AUC) of leniolisib in pediatric patients (aged 4 to 11 years) with APDS | From baseline to end of 12 weeks of treatment
  Population pharmacokinetics (popPK) model that describes the appropriate covariates (eg, body weight and age) that influence leniolisib PK in pediatric patients.
Part I: To assess the maximum concentration (Cmax) of leniolisib in pediatric patients (aged 4 to 11 years) with APDS | From baseline to end of 12 weeks of treatment
  Population pharmacokinetics (popPK) model that describes the appropriate covariates (eg, body weight and age) that influence leniolisib PK in pediatric patients.
Part I: To assess the time to maximum concentration (Tmax) of leniolisib in pediatric patients (aged 4 to 11 years) with APDS | From baseline to end of 12 weeks of treatment
  Population pharmacokinetics (popPK) model that describes the appropriate covariates (eg, body weight and age) that influence leniolisib PK in pediatric patients.
Part II: Changes from baseline for Reduction in lymphadenopathy as measured by MRI or low-dose CT | Day 85 to through study completion, an average of 1 year
  Parameters for reduction in lymphadenopathy as a key secondary endpoint of Part II may include 3D volume of index and measurable non-index lesions selected as per the Cheson methodology. Summary statistics will be provided by visit. Arithmetic mean with SD of absolute values and change from baseline values may be plotted across time.
Part II: Changes from baseline for Reduction in lymphadenopathy as measured by MRI or low-dose CT | Day 85 to through study completion, an average of 1 year
  Parameters for reduction in 3D volume and bi-dimensional or 3D sizes of spleen, where appropriate. Summary statistics will be provided by visit. Arithmetic mean with SD of absolute values and change from baseline values may be plotted across time.
Part II: Changes from baseline for Reduction in lymphadenopathy as measured by MRI or low-dose CT | Day 85 to through study completion, an average of 1 year
  Parameters for reduction in 3D volume and bi-dimensional or 3D sizes of liver, where appropriate. Summary statistics will be provided by visit. Arithmetic mean with SD of absolute values and change from baseline values may be plotted across time.
Part I and II: Key secondary efficacy outcomes for Part I include incidence of infections and use of antibiotics. | Part I: Baseline to Day 85 Part II: through study completion, an average of 1 year
  The number and percentage of patients with infections, and the total number of infections will be summarized. The number and percentage of antibiotics taken will be presented along with number of patients for Part I. Use of immunoglobulin replacement therapy over time will be summarized.
Part I and II: Pediatric Quality of Life Inventory (PedsQLTM) Parent Report for Children Questionnaire 4.0 Generic Core Scales | Part I: Baseline, Day 29, 57, & 85 Part II: through study completion, an average of 1 year
  To assess the ability of leniolisib to modify health related quality of life in pediatric patients with APDS. The unabbreviated scale title is SCALING AND SCORING OF THE PedsQL. The minimum and maximum values; are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Higher scores indicate better HRQOL.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Standford, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - National Institutes of Health, Bethesda, Maryland
- Necker Hospital Paris, Paris, France
- Japan (2):
  - Kyoto University Hospital, Kyoto
  - Institute of Science Tokyo Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No